CLINICAL TRIAL: NCT02638792
Title: Internet-Based Exposure Therapy Vs. Stress-Management Training for Worry: A Randomized Controlled Trial
Brief Title: Internet-Based Exposure Therapy Vs. Stress-Management Training for Worry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, PhD, Lic. psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REPN 2015/1698-31/1
Record Dates: First submitted 2015-12-19; First posted 2015-12-23 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Excessive Worry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Internet-based exposure therapy (Experimental): The internet-based exposure therapy (I-ET) group receives a ten-week Internet-based CBT treatment, which is an extended version of the self-help book "Sluta älta och grubbla med kognitiv beteendeterapi" (How to quit worrying and ruminating with Cognitive behavior therapy) by licensed psychologist Olle Wadström (2007). The main focus of the book is to expose to the frightening word/image and refrain from using neutralizing thoughts. This is supposed to lead to the extinction of upsetting words/images.
  Interventions: Behavioral: Internet-based exposure therapy (I-ET)
- Internet-based stress management therapy (Active Comparator): The I-SMT group receives a ten-week Internet-based CBT treatment focused on stress and how to manage stressful situations. This protocol is based on current evidence based recommendations for worry and has shown to be effective when delivered via the internet for irritable bowel syndrome and hypochondric worries.
  Interventions: Behavioral: Internet-based stress management therapy
- Waitlist (No Intervention): When the active treatment groups have finished treatment (W11), the WL group will be able to start active treatment and be assessed at post-treatment, and 4, 12 months later using the same questionnaires as the treatment group. The participants will be able to choose which treatment they receive i.e. no randomization.

INTERVENTIONS:
Behavioral: Internet-based exposure therapy (I-ET) — The internet-based exposure therapy (I-ET) group receives a ten-week Internet-based CBT treatment, which is an extended version of the self-help book "Sluta älta och grubbla med kognitiv beteendeterapi" (How to quit worrying and ruminating with Cognitive behavior therapy) by licensed psychologist Olle Wadström (2007). The main focus of the book is to expose to the frightening word/image and refrain from using neutralizing thoughts. This is supposed to lead to the extinction of upsetting words/images.
  Arms: Internet-based exposure therapy
Behavioral: Internet-based stress management therapy — The I-SMT group receives a ten-week Internet-based CBT treatment focused on stress and how to manage stressful situations. This protocol is based on current evidence based recommendations for worry and has shown to be effective when delivered via the internet for irritable bowel syndrome and hypochondric worries.
  Arms: Internet-based stress management therapy

SUMMARY:
The purpose of this study is to examine if an internet-based exposure therapy is more effective in reducing excessive worry amongst patients who suffer from this problem than is internet-based stress management training.

DETAILED DESCRIPTION:
Trial Objectives: Primary objective is to investigate whether an Internet-based exposure therapy can reduce the degree of excessive worry to a significantly greater extent than Internet-based stress-management training. The secondary objective is to a) investigate the cost-effectiveness of this treatment b) to study if any variables could moderate/mediate the treatment outcome, c) and to investigate the importance of sudden gains for the treatment outcome

Trial Design: Randomized controlled trial with an active control and a waitlist control, who also will recieve treatment after the first group has finished.

Duration: Ten weeks

Primary Endpoint:

Difference in worry symptoms between the treatment groups at week 10. Long term follow-up is also investigated (baseline to 4-months after treatment completion and baseline to 12-months after treatment completion).

Efficacy Parameters: Penn State Worry Questionnaire (PSWQ)

Safety Parameters: Adverse Events is assessed via the internet.

Description of Trial Subjects: Patients > 18 years old with a PSWQ score more than 56 points

Number of Subjects: 300

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* ≥ 18 years
* Situated in Sweden
* Informed consent
* PSWQ score more than 56 points

Exclusion Criteria:

* Substance dependence during the last six months
* Post traumatic stress disorder, bipolar disorder or psychosis
* Symptoms better explained by axis 2 diagnosis (e.g. autism or borderline personality disorder)
* MADRS-S score above 25 points
* Psychotropic medication changes within two months prior to treatment that could affect target symptoms.
* Received exposure based CBT for pathological worry the last 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | week 0, week 10 (weekly measurements), at 4 months follow up, 12 months follow up.
  Change in worry from baseline to Week 10 and at 4- and 12 months after treatment has ended.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale (MADRS-S) | Week 0, Week 10, 4 and 12 months follow-up
  Change in depression from baseline to Week 10 and at 4- and 12 months after treatment has ended.
Euroqol, EQ-5D | Week 0, Week 10, 4 and 12 months follow-up
  Change in general health from baseline to Week 10 and at 4- and 12 months after treatment has ended
Cognitive Avoidance Questionnaire (CAQ) | Week 0, Week 10, at 4 and 12 months follow up and weekly during treatment
  Change in cognitive avoidance from baseline to Week 10, at 4- and 12 after treatment has ended, and weekly during treatment
Intolerance of uncertainty scale | Week 0, Week 10, at 4 and 12 months follow-up, and weekly during treatment
  Change in thought control efforts from baseline to Week 10, at 4- and 12 months after treatment has ended, and weekly during treatment
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | Week 0, Week 10, 4 and 12 months follow-up
  Change in economic costs from baseline to Week 10 and at 4- and 12 months after treatment has ended
Brunnsviken Quality of Life Questionnaire (BBQ) | Week 0, Week 10, 4 and 12 months follow-up
  Change in self-perceived quality of life from baseline to week 10 and at 4 and 12 months after treatment has ended
Thought supression subscale of the Cognitive Avoidance Questionnaire (CAQ) | Week 0 - Week 10 (weekly measurements)
  Weekly change in thought supression from baseline to Week 10
The self-regulation subscale of the Multidimensional Assessment of Interoceptive Awareness | Week 0 - Week 10 (weekly measurements)
  Weekly change in self-regulation from baseline to Week 10
Patient Health Questionnaire-2 | Week 0 - Week 10 (weekly measurements)
  Weekly change in depressive symptom from baseline to Week 10
Adverse Events | Week 3, week 8, week 10, 4 and 12 months follow-up
  Number of adverse events from baseline to Week 10 and at 4 and 12 months

OTHER OUTCOMES:
Treatment credibility scale | Week 2
  Investigate if both conditions have equal credibility in order to rule out placebo
Working alliance scale | Week 5
  Investigate if both conditions have equal working alliance in order to rule out non-specific factors

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Andersson, PhD, Psych., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Intitutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No